CLINICAL TRIAL: NCT01251016
Title: Changes in Gene Expression of Intestinal Tissue From Type 2 Diabetes Patients Submitted to Roux-en-Y Gastric Bypass
Brief Title: Effect of Bariatric Surgery on Gut Hormones Production and Cure of Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Pennington Biomedical Research Center (Other); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Dan Linetzky Waitzberg, Associate Professor, University of Sao Paulo
Other Study IDs: CAPPesq 1011/09
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Surgery
Keywords: Type 2 diabetes mellitus; Y-Roux gastric bypass; Gut hormones; Gene expression; Surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a relevant public health problem and obesity has been associated as the major risk factor. Roux-en-Y gastric bypass is an effective method to treat severe obesity, and its metabolic benefits can lead to early and complete remission of T2DM, even before a considerable weight loss. We have hypothesized that intestinal anatomic changes may change intestinal genes expression related to glycemic control. The knowledge of mechanisms mediating the glycemic control after Roux-en-Y gastric bypass and it site of action in bowel may eventually help to develop alternative, less invasive and safer surgery for the treatment of T2DM, as well as drug development for the newly targets identified.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes mellitus (T2DM) diagnosis Duration of T2DM >5 years Use of oral antidiabetic agents Body Mass Index >40 kg/m2 Candidates to Roux-en-Y gastric bypass

Exclusion Criteria:

Type 1 diabetes mellitus or non-diabetics Use of insulin Thyroid diseases Candidate to other surgery technique Body Mass Index <40 kg/m2 Presence of bacterium H. Pylori

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Severe obese patients with T2DM candidates to Roux-en-Y gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Patient Selection | 2013
  10 patients fully completed with all biological samples colected in the preoperative and postoperative periods (gastrointestinal tissue). RNA extraction of gastrointestinal samples is being performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinics Hospital of the University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lemos GO, Torrinhas RS, Machado NM, Waitzberg DL. Changes in Plasma Sphingolipid Metabolites Following Roux-En-Y Gastric Bypass in Women With Obesity and Type 2 Diabetes: A Pilot Metabolomic Cohort Study. Lipids. 2025 Nov 12. doi: 10.1002/lipd.70019. Online ahead of print. PMID 41224249
- [Derived] Garla P, Sala P, Torrinhas RSM, Machado NM, Fonseca DC, da Silva MM, Ravacci GR, Belarmino G, Ishida RK, Guarda IFMS, de Moura EGH, Sakai P, Santo MA, da Silva IDCG, Pereira CCA, Heymsfield S, Correa-Giannella MLC, Calder PC, Waitzberg DL. Reduced intestinal FADS1 gene expression and plasma omega-3 fatty acids following Roux-en-Y gastric bypass. Clin Nutr. 2019 Jun;38(3):1280-1288. doi: 10.1016/j.clnu.2018.05.011. Epub 2018 May 29. PMID 30459098
- [Derived] Sala P, Torrinhas RS, Fonseca DC, Heymsfield S, Giannella-Neto D, Waitzberg DL. Type 2 Diabetes Remission After Roux-en-Y Gastric Bypass: Evidence for Increased Expression of Jejunal Genes Encoding Regenerating Pancreatic Islet-Derived Proteins as a Potential Mechanism. Obes Surg. 2017 Apr;27(4):1123-1127. doi: 10.1007/s11695-017-2602-0. PMID 28213664
- [Derived] Silva MM, Sala PC, Cardinelli CS, Torrinhas RS, Waitzberg DL. Comparison of Virtual Nutri Plus(R) and Dietpro 5i(R) software systems for the assessment of nutrient intake before and after Roux-en-Y gastric bypass. Clinics (Sao Paulo). 2014 Nov;69(11):714-22. doi: 10.6061/clinics/2014(11)02. PMID 25518027